CLINICAL TRIAL: NCT01430169
Title: A Phase 2, Open-Label Study to Assess the Pharmacokinetics of a Single Treatment Cycle of AA4500 0.58 mg in Men With Peyronie's Disease
Brief Title: Pharmacokinetics of a Single Treatment Cycle of AA4500 0.58 mg in Men With Peyronie's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUX-CC-805
Record Dates: First submitted 2011-09-06; First posted 2011-09-08 (Estimated); Results first posted 2015-05-06 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Peyronie's Disease
Keywords: Xiaflex; Xiapex; Collagenase clostridium histolyticum
MeSH Terms: conditions — Penile Induration | interventions — Microbial Collagenase; xiapex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AA4500 (Experimental): collagenase clostridium histolyticum (AA4500) contains purified collagenase AA4500 (clostridium histolyticum) consisting of two microbial collagenases in a defined mass ratio, Collagenase AUX-I and Collagenase AUX-II, which are isolated and purified from the fermentation of Clostridium histolyticum bacteria.
  2 injections of AA4500 0.58 mg were administered 24 hours apart.
  Interventions: Biological: AA4500

INTERVENTIONS:
Biological: AA4500 — Two injections of AA4500 0.58 mg 24 hours apart
  Other Names: XIAFLEX, XIAPEX

SUMMARY:
This study is a Phase 2, open-label study to assess the pharmacokinetics (PK) and safety of AA4500 0.58 mg in men with Peyronie's disease. Subjects will be screened for study eligibility within 21 days before the initial injection of study drug. Two injections will be administered 24 hours apart.

Subjects will be admitted to the study unit the day before the first injection of AA4500 (Day -1) and will remain in the study unit until after the PK sample is collected after investigator penile plaque modeling on Day 3. Subjects will return to the study unit on Day 4, Day 8, and Day 29 for follow-up pharmacokinetic and safety assessments.Pharmacokinetic plasma samples will be collected at predetermined time points before (15 minutes pre-injection) and after each injection on Day 1 and Day 2 (5,10, 20, 30 minutes and 1,2,3,4,8,12 hours after), and on Days 3, 4, 8, and 29.Plasma levels for AUX-I (clostridial type I collagenase) and AUX-II (clostridial type II collagenase) will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Be a male and be ≥ 18 years of age
2. Be in a stable relationship with a female partner/spouse for at least 3 months before screening and be willing to have vaginal intercourse with that partner/spouse
3. Have symptom(s) of Peyronie's disease for at least 12 months before the first dose of study drug and have evidence of stable disease as determined by the investigator
4. Have penile curvature of at least 30° in the dorsal, lateral, or dorsal/lateral plane at screening. It must be possible to delineate the single plane of maximal curvature for evaluation during the study
5. Be judged to be in good health, based upon the results of a medical history, physical examination, and laboratory profile
6. Voluntarily sign and date an informed consent agreement approved by the Institutional Review Board/Independent Ethics Committee (IRB/IEC). The subject must also sign an authorization form to allow disclosure of his protected health information (PHI). The PHI authorization form and informed consent form may be an integrated form or may be separate forms depending on the institution
7. Be able to read, complete and understand the various rating instruments in English

Exclusion Criteria:

A subject will be excluded from study participation if he:

1. Has a penile curvature of less than 30° or greater than 90° at the screening visit
2. Has any of the following conditions:

   Chordee in the presence or absence of hypospadias; Thrombosis of the dorsal penile artery or vein; Infiltration by a benign or malignant mass resulting in penile curvature; Infiltration by an infectious agent, such as lymphogranuloma venereum; Ventral curvature from any cause; Presence of an active sexually transmitted disease; Known active hepatitis B or C; Known immune deficiency disease or be positive for human immunodeficiency virus (HIV)
3. Has previously undergone surgery for Peyronie's disease
4. Fails to have an erection which in the opinion of the investigator is sufficient to accurately measure the subject's penile deformity after administration of an appropriate pharmacological stimulant (eg, prostaglandin E1 or trimix)
5. Has a calcified plaque as evident by appropriate radiographic evaluation, penile x-ray or penile ultrasound that would prevent proper injection of study medication. Non-contiguous stippling of calcium is acceptable for inclusion provided the calcium deposit does not interfere with the injection of AA4500 into the plaque
6. Has an isolated hourglass deformity of the penis (curvature caused by a plaque that is noncontiguous with the hourglass deformity may be treated)
7. Has the plaque causing curvature of the penis located proximal to the base of the penis, so that the injection of a local anesthetic would interfere with the injection of AA4500 into the plaque
8. Has previously received alternative medical therapies for Peyronie's disease administered by the intralesional route (including, but not limited to, steroids, verapamil, and the naturally occurring low molecular weight protein, interferon-α2b) within 3 months before the first dose of study drug or plans to use any of these medical therapies at any time during the study
9. Has received alternative medical therapies for Peyronie's disease administered by the oral (including, but not limited to, vitamin E [>500 U], potassium aminobenzoate [Potaba], tamoxifen, colchicine, pentoxifylline, over-the-counter erectile dysfunction medications, or steroidal anti-inflammatory drugs) or topical routes (including, but not limited to, verapamil applied as a cream) within 3 months before the first dose of study drug or plans to use any of these medical therapies at any time during the study
10. Has had extracorporeal shock wave therapy (ESWT) for the correction of Peyronie's disease within the 6- month period before screening or plans to have ESWT at any time during the study
11. Has used any mechanical type device for correction of Peyronie's disease within the 2-week period before screening or plans to use any these devices at any time during the study
12. Has used a mechanical device to induce a passive erection within the 2-week period before screening or plans to use any of these devices at any time during the study
13. Has significant erectile dysfunction that has failed to respond to oral treatment with phosphodiesterase type 5 (PDE5) inhibitors
14. Has a penile Duplex Doppler ultrasound evaluation at screening that shows compromised penile hemodynamics that in the opinion of the investigator is clinically significant
15. Has uncontrolled hypertension, as determined by the investigator
16. Has a known recent history of stroke, bleeding, or other significant medical condition, which in the investigator's opinion would make the subject unsuitable for enrollment in the study
17. Is unwilling or unable to cooperate with the requirements of the study including completion of all scheduled study visits
18. Has received an investigational drug or treatment within 30 days before the first dose of study drug
19. Has a known systemic allergy to collagenase or any other excipient of AA4500
20. Has a known allergy or contraindication to any concomitant medication required as per the protocol
21. Has received anticoagulant medication (except for ≤ 165 mg aspirin daily or ≤ 800 mg of over-the-counter NSAIDS daily) during the 7 days before the first dose of study drug
22. Has received tetracycline, doxycycline, or other tetracycline derivatives within 5 days before the first dose of study drug or plans to use any of these drugs at any time during the study
23. Has received any collagenase treatments within 30 days of the first dose of study drug
24. Has, at any time, received AA4500 for the treatment of Peyronie's disease
25. Has a positive alcohol breath test or positive urine drug screen for amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, and/or propoxyphene at screening and/or on Day -1
26. Has a 12-lead electrocardiogram (ECG) finding that is outside 'normal limits' or interpreted as 'abnormal, clinically significant', as determined by the physician

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J. Kaufman, MD, Study Director — Auxilium Pharmaceuticals, Inc.
Locations (1):
- Martin Gelbard, MD Inc., Burbank, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- AA4500: collagenase clostridium histolyticum
  AA4500: Two injections of AA4500 0.58 mg (First Injection is administered on Day 1 and the second Injection is administered on Day 2)
Period: Overall Study
Arm/Group | AA4500
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- AA4500: collagenase clostridium histolyticum
  AA4500: Two injections of AA4500 0.58 mg
Arm/Group | AA4500
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (8.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: AUX-I Cmax After Injection 1
Description: Maximum AUX-I (clostridial type I collagenase) enzyme concentration from pre-injection to 24 hours after Injection 1. AUX-I plasma concentrations were determined with a validated enzyme-linked immunosorbent assay (ELISA).
Time Frame: 15 minutes before Injection 1 (0 hour for Injection 1); 5, 10, 20, and 30 minutes after Injection 1; 1, 2, 4, 8, and 12 hours after Injection 1; 15 minutes before Injection 2 (24 hours after Injection 1)
Population: Pharmacokinetic (PK) population (N=19). Two subjects were excluded from the analysis due to bioanalytical reasons (ELISA interference)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AA4500
Number analyzed (Participants) | 17
ng/mL | 12.6 (8.3)

2. Primary Outcome: AUX-II Cmax After Injection 1
Description: Maximum AUX-II (clostridium Type II collagenase) enzyme concentration from pre-injection to 24 hours after Injection 1. AUX-II plasma concentrations were determined with a validated enzyme-linked immunosorbent assay (ELISA).
Time Frame: as for outcome 1
Population: Pharmacokinetic (PK) population (N=19).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AA4500
Number analyzed (Participants) | 19
ng/mL | 15.1 (19.2)

3. Primary Outcome: AUX-I AUC0-tlast After Injection 1
Description: Area under the curve from pre-injection to tlast within 24 hours after the Injection 1, where tlast is time to last time with a quantifiable concentration of the enzyme AUX-I. AUX-I plasma concentrations were determined with a validated enzyme-linked immunosorbent assay (ELISA).
Time Frame: as for outcome 1
Population: Pharmacokinetic population (N=19). Two subjects were excluded from the analysis due to bioanalytical reasons (ELISA interference)
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | AA4500
Number analyzed (Participants) | 17
ng*h/mL | 3.1 (2.1)

4. Primary Outcome: AUX-II AUC0-tlast After Injection 1
Description: Area under the curve from pre-injection to tlast within 24 hours after the Injection 1, where tlast is time to last time with a quantifiable concentration of the enzyme AUX-II. AUX-II plasma concentrations were determined with a validated enzyme-linked immunosorbent assay (ELISA).
Time Frame: as for outcome 1
Population: Pharmacokinetic (PK) population (N=19)
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | AA4500
Number analyzed (Participants) | 19
ng*h/mL | 2.2 (3.9)

5. Primary Outcome: AUX-I Tmax After Injection 1
Description: Time to maximum AUX-I enzyme concentration. AUX-I plasma concentrations were determined with a validated enzyme-linked immunosorbent assay (ELISA).
Time Frame: as for outcome 1
Population: Pharmacokinetic (PK) population (N=19). For 3 subjects Tmax was considered missing if concentration was BLQ for all time points at that injection and 2 subjects were excluded from the analysis due to bioanalytical reasons (ELISA interference)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | AA4500
Number analyzed (Participants) | 14
hours | 0.15 (0.09)

6. Primary Outcome: AUX-II Tmax After Injection 1
Description: Time to maximum AUX-II enzyme concentration. AUX-II plasma concentrations were determined with a validated enzyme-linked immunosorbent assay (ELISA).
Time Frame: as for outcome 1
Population: Pharmacokinetic (PK) population (N=19) One subject was excluded from AUX-II PK analyses due to insufficient quantities of plasma for bioanalysis. Of the 38 AUX-II profiles, 23 had no quantifiable plasma concentrations at any time point through 24 hours post injection.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | AA4500
Number analyzed (Participants) | 8
hours | 0.16 (0.08)

7. Primary Outcome: AUX-I Cmax After Injection 2
Description: Maximum AUX-I enzyme concentration from zero to 24 hours after Injection 2.AUX-I plasma concentrations were determined with a validated enzyme-linked immunosorbent assay (ELISA).
Time Frame: 15 minutes before Injection 2 (24 hours after Injection 1 or 0 hour for Injection 2); 5, 10, 20, and 30 minutes after Injection 2; 1, 2, 4, 8, and 12 hours after Injection 2; Day 3 (24 hours after Injection 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AA4500
Number analyzed (Participants) | 17
ng/mL | 12.2 (9.1)

8. Primary Outcome: AUX-II Cmax After Injection 2
Description: Maximum AUX-II enzyme concentration from zero to 24 hours after Injection 2. AUX-II plasma concentrations were determined with a validated enzyme-linked immunosorbent assay (ELISA).
Time Frame: as for outcome 7
Population: Pharmacokinetic (PK) population (N=19)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AA4500
Number analyzed (Participants) | 19
ng/mL | 16.1 (23.2)

9. Primary Outcome: AUX-I AUC0-tlast After Injection 2
Description: Area under the curve from zero to tlast within 24 hours after the Injection 2, where tlast is time to last time with a quantifiable concentration of the enzyme AUX-I. AUX-I plasma concentrations were determined with a validated enzyme-linked immunosorbent assay (ELISA).
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | AA4500
Number analyzed (Participants) | 17
ng*h/mL | 2.4 (2.3)

10. Primary Outcome: AUX-II AUC0-tlast After Injection 2
Description: Area under the curve from zero to tlast within 24 hours after the Injection 2, where tlast is time to last time with a quantifiable concentration of the enzyme AUX-II. AUX-II plasma concentrations were determined with a validated enzyme-linked immunosorbent assay (ELISA).
Time Frame: as for outcome 7
Population: Pharmacokinetic (PK) population (N=19)
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | AA4500
Number analyzed (Participants) | 19
ng*h/mL | 2.3 (4.1)

11. Primary Outcome: AUX-I Tmax After Injection 2
Description: as for outcome 5
Time Frame: as for outcome 7
Population: Pharmacokinetic (PK) population (N=19). In addition, 2 subjects have been excluded from the analysis due to ELISA interference.
  Of the 38 AUX-I profiles, 7 had no quantifiable plasma concentrations through 24 hours post injection.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | AA4500
Number analyzed (Participants) | 13
hour | 0.11 (0.07)

12. Primary Outcome: AUX-II Tmax After Injection 2
Description: as for outcome 6
Time Frame: as for outcome 7
Population: Pharmacokinetic (PK) population (N=19) In addition, 2 subjects have been excluded from the analysis due to ELISA interference. Of the 38 AUX-II profiles,23 had no quantifiable plasma concentrations at any time point through 24 hours post injection.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | AA4500
Number analyzed (Participants) | 7
hours | 0.12 (0.09)

ADVERSE EVENTS:
Time Frame: 28 days after the first injection
Arm/Group | AA4500
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 (N=20)
Penile haemorrhage (Reproductive system and breast disorders) | 19 (23) — Verbatim term is penile ecchymosis
Injection site pain (General disorders) | 15 (15)
Procedural pain (Injury, poisoning and procedural complications) | 9 (10)
Penile swelling (Reproductive system and breast disorders) | 6 (6)
Painful erection (Reproductive system and breast disorders) | 4 (4)
Penile pain (Reproductive system and breast disorders) | 4 (5)
Post procedural discomfort (Injury, poisoning and procedural complications) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Injection site haemorrhage (General disorders) | 1 (1)
Penile blister (Reproductive system and breast disorders) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other